CLINICAL TRIAL: NCT00611624
Title: A Phase II Trial of Mammosite Breast Brachytherapy Optimization in the Treatment of Stage 0, I and II Breast Carcinoma
Brief Title: Mammosite Breast Brachytherapy Optimization in the Treatment of Breast Carcinoma
Acronym: Mammosite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0601000957
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-02

CONDITIONS: Breast Neoplasms
Keywords: MammoSite; brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Five Days of Mammosite Therapy (Experimental): Five Days of Mammosite Therapy (Radiotherapy)
  Interventions: Radiation: Mammosite brachytherapy radiation

INTERVENTIONS:
Radiation: Mammosite brachytherapy radiation — Treatment using MammoSite will begin within five days of placement of the catheter. Only high dose rate (HDR) with Ir-192 treatment is allowed. The balloon will remain inflated throughout the treatment course. A total of 34 Gy will be prescribed to an approximate 1 cm radial distance from the balloon surface. Two fractions per day, each of 3.4 Gy, separated by at least 6 hours, given on 5 treatment days (over a period of 5 to 10 days), will sum to 10 fractions and 34 Gy.

SUMMARY:
The purpose of this study is to determine if Mammosite Catheter optimization using multiple dwell position delivery decreases skin toxicity over historically reported skin toxicity with the single dwell delivery method.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have a signed an approved consent form conforming with institutional guidelines.
* Patient must be > 50 years old.
* The patient should have a life expectancy of at least two years.
* The patient must have stage 0 , I , or II breast cancer. If stage IIA, the tumor size must be 3 cm or less and the patients must be node negative.
* On histological examination, the tumor must be DCIS or invasive adenocarcinoma of the breast.
* Surgical treatment of the breast must have been lumpectomy. The margins of the resected specimen must be histologically free of tumor (>2mm, DCIS and invasive). Re-excision of surgical margins is permitted.
* Gross disease must be unifocal with pathologic (invasive and/or DCIS) tumor size 3 cm or less. (Patients with microscopic multifocality are eligible as long as total pathologic tumor size is 3 cm or less.)
* Patients with invasive breast cancer are required to have axillary staging which can include sentinel node biopsy alone (if negative), sentinel node biopsy followed by axillary dissection or sampling with a minimum total of 6 axillary nodes or axillary dissection alone (with a minimum of 6 axillary nodes). (Axillary staging is NOT required for patients with DCIS.)
* The patient must have the MammoSite catheter placed within 4 weeks or 28 days of the final surgery for their breast cancer (lumpectomy, re-excision of margins, or axillary staging procedure). Placement of a spacer for the MammoSite catheter is permitted at their final surgery.
* Patients with a history of non-ipsilateral breast malignancies are eligible if they have been disease-free for 2 or more years prior to randomization. Patients with the following cancers are eligible even if diagnosed and treated within the past 2 years: carcinoma in situ of the cervix, colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin. Patients with a prior diagnosis of ipsilateral breast cancer are ineligible.
* Chemotherapy is permitted if planned for >2 weeks after removal of Mammosite catheter.
* Patient must be ineligible or have refused enrollment on the randomized trial RTOG (Radiation Therapy Oncology Group) 0413.

Exclusion Criteria:

* Men are not eligible for this study.
* T2 (>3.0 cm), T3, node positive, stage III or IV breast cancer.
* Any positive axillary nodes.
* Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular or internal mammary nodes, unless biopsy proven to be negative for tumor.
* Suspicious microcalcifications, densities or palpable abnormalities in either breast unless biopsy proven to be benign.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma in more than one quadrant or separated by more than 3 centimeters.
* Paget's disease of the nipple.
* History of invasive breast cancer or DCIS in the same breast.
* Surgical margins that cannot be microscopically assessed or are less then 2 mm.
* Collagen vascular disease, specifically dermatomyositis with a creatine phosphokinase (CPK) level above normal or with an active skin rash, systemic lupus erythematosis or scleroderma.
* Pregnancy or lactation at the time of proposed radiation. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Patients with coexisting medical conditions in whom life expectancy is < 2 years.
* Patients with skin involvement, regardless of tumor size.
* Patients for whom treatment with the MammoSite catheter is not feasible, such as those with too little breast tissue between the skin and the catheter (as determined by distance of dose calculations).

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Weidhaas, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Five Days of Mammosite Therapy
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Five Days of Mammosite Therapy
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Tumor Stage [Count of Participants; unit: Participants] — Breast cancer tumor size was determined prior to study inclusion. Tis is Carcinoma in situ. T1 tumors are 2 cm or smaller. T1mi is Tumor ≤ 1 0.1cm in greatest dimension. T1a - T1c is ordered smallest to largest (all under 2 cm).
  Participants
    Tis | 4
    T1mi | 1
    T1a | 2
    T1b | 10
    T1c | 11
Histology [Count of Participants; unit: Participants]
  Ductal carcinoma in situ (DCIS) | 4
  Invasive ductal carcinoma | 19
  Invasive lobular carcinoma | 3
  Invasive tubulolobular carcinoma | 1
  Invasive cribriform carcinoma | 1
Lymph node evaluation [Count of Participants; unit: Participants] — Only those with invasive disease were counted. Population: n = 24
  Participants
    number analyzed (Participants) | 24
    Sentinel lymph node | 24
    Axillary lymph node dissection | 0
Size of invasive component [Median (Full Range); unit: centimeters (cm)] | 1.0 [0.1 to 2.0]
Size of in situ component [Median (Full Range); unit: centimeters (cm)] | 0.8 [0 to 2.8]
Size of in situ component (DCIS patients) [Median (Full Range); unit: centimeters (cm)] — Population: This was only measured in DCIS patients (n=4).
  centimeters (cm)
    number analyzed (Participants) | 4
    (all) | 0.8 [0.3 to 2.2]
estrogen receptor (ER) [Count of Participants; unit: Participants]
  positive | 28
  negative | 0
progesterone receptor (PR) [Count of Participants; unit: Participants]
  positive | 24
  negative | 4
HER2/neu status (invasive disease only) [Count of Participants; unit: Participants] — Population: Only counted in those with invasive disease (n=24).
  Participants
    number analyzed (Participants) | 24
    positive | 0
    negative | 24
lymphovascular space invasion (LVSI) [Count of Participants; unit: Participants]
  yes | 0
  no | 28

OUTCOME MEASURES:

1. Primary Outcome: Skin Toxicity the First Year Following Treatment With the Multiple Dwell Mammosite Delivery Method.
Description: Evaluation of skin toxicity the first year following treatment with the multiple dwell Mammosite delivery method. The number of participants with a grade 2 skin toxicity (or higher) at 1 year follow up are reported. Radiation Therapy Oncology Group (RTOG) and the European organization for research and treatment of cancer (EORTC) Late Radiation Morbidity Scoring Schema were used to assess toxicity.
Time Frame: one year
Population: 26 participants completed the 1 year assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Five Days of Mammosite Therapy
Number analyzed (Participants) | 26
Participants
  Grade 2 Toxicity | 2
  Grade 3 Toxicity | 0
  Grade 4 Toxicity | 0
  Grade 5 Toxicity | 0
  Did not experience >= Grade 2 Toxicity | 24

2. Secondary Outcome: Information of Treatment Parameters in Order to Define Parameters Most Predictive of Skin Toxicity
Description: These data were not collected and were not summarized in this study. Results are not available.
Time Frame: Upon completion of study
Groups:
- Patient Characteristics: Twenty-eight women in total were enrolled and had been treated on this trial at the time of analysis (12 additional patients accrued after the initial phase of 16 patients).
Arm/Group | Patient Characteristics
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Five Days of Mammosite Therapy
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 13/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Five Days of Mammosite Therapy (N=28)
Pain (General disorders) | 2 (2)
Fibrosis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Telangiectasia (Vascular disorders) | 2 (2)
Skin (Skin and subcutaneous tissue disorders) | 2 (2) — All skin related issues

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes